CLINICAL TRIAL: NCT01789463
Title: Physiotherapy Versus Self Rehabilitation After Shoulder Dilatation for Primary Idiopathic Capsulitis
Brief Title: Physiotherapy and Capsulitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/03
Record Dates: First submitted 2013-01-10; First posted 2013-02-12 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self rehabilitation (Active Comparator): Self rehabilitation
  Interventions: Other: Self rehabilitation
- Self rehabilitation plus physiotherapy (Experimental): Self rehabilitation plus physiotherapy
  Interventions: Other: Self rehabilitation plus physiotherapy

INTERVENTIONS:
Other: Self rehabilitation
  Arms: Self rehabilitation
Other: Self rehabilitation plus physiotherapy
  Arms: Self rehabilitation plus physiotherapy

SUMMARY:
Multicenter randomised study, on parallel groups to compare recovery of functional amplitude following shoulder dilatation with auto rehabilitation in one group and physiotherapy in the other group.

ELIGIBILITY:
Inclusion Criteria:

* Primary idiopathic phase 2 capsulitis
* Diagnosis of capsulitis confirmed by shoulder dilatation
* Patients between 18 and 70 years of age
* Exclusion Criteria:
* Secondary capsulitis
* Shoulder pain of other etiology
* Cognitive disorders
* Patients less than 18 years, and more than 70 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Function of the shoulder joint (Score de Constant) | 12 months post shoulder dilatation

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (at evening, rest, and at movement) | 12 months post shoulder dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Bernard BOISAUBERT, MD, Study Chair — Hôpital FOCH 40, rue Worth 92150 Suresnes; Louis FRANCESCHI, MD, Principal Investigator — IMM - 42, boulevard Jourdan 75014 Paris
Locations (1):
- Hôpital FOCH, Suresnes, France